CLINICAL TRIAL: NCT02380950
Title: Effect of Moderate Alcohol Consumption to Cognitive Functioning After Roux-en Y Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: eSwiss Medical & Surgical Center (Other)
Responsible Party: Principal Investigator, Bernd Schultes, Prof. Dr. med. Bernd Schultes, eSwiss Medical & Surgical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EKSG 13/046
Record Dates: First submitted 2015-02-19; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Bariatric Surgery; Alcohol Consumption; Cognitive Function
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

ARMS (1):
- 250 ml alcohol consumption (Other): Each participant had to drink 250 ml white wine. Directly before, 10-30 min after and 45-65 min after wine consumption cognitive functions were tested by test battery for attentional performance (TAP) from Zimmermann and Fimm. During the whole examination breath-alcohol-contents (BACs) were measured every 5 minutes with breathalyser "Dräger Alcotest 7510".
  Interventions: Behavioral: 250 ml alcohol consumption

INTERVENTIONS:
Behavioral: 250 ml alcohol consumption — Each participant had to drink 250 ml white wine. Directly before, 10-30 min after and 45-65 min after wine consumption cognitive functions were tested by test battery for attentional performance (TAP) from Zimmermann and Fimm. During the whole examination breath-alcohol-contents (BACs) were measured every 5 minutes with breathalyser "Dräger Alcotest 7510".

SUMMARY:
Objectives: Alcohol metabolism is changed in gastric bypass patients, leading to faster resorption and higher alcohol peak concentrations in blood. Because of stronger alcohol effects after gastric bypass we suggest that also general cognitive function is stronger impaired.

Materials and Methods: We included 28 females (12 gastric bypass patients, 8 obese and 8 normal weight subjects) in the study. Each participant had to drink 250 ml white wine. Directly before, 10-30 min after and 45-65 min after wine consumption cognitive functions were tested by test battery for attentional performance (TAP) from Zimmermann and Fimm. During the whole examination breath-alcohol-contents (BACs) were measured every 5 minutes with breathalyser "Dräger Alcotest 7510".

ELIGIBILITY:
Inclusion Criteria:

Gastric bypass group:

* women
* preOP BMI >35 kg/m²
* time since bariatric surgery > 1 year
* age 18-60 years
* moderate drinking habits

obese group:

* women
* BMI >35 kg/m²
* age 18-60 years
* moderate drinking habits

normal weight group:

* women
* BMI 18.5 - 25 kg/m²
* age 18-60 years
* moderate drinking habits

Exclusion Criteria:

* men
* patient does not drink wine
* usage of psychotropic drugs
* alcoholic
* pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in reaction time after alcohol consumption | Change measures (baseline, 10 min, 45 min)